CLINICAL TRIAL: NCT02650115
Title: Evaluation of the Involvement of the Intestinal Microbiota and Choline Deficiency in the Severity of Chronic Liver Disease Explored by Analyzing Collection of Biological Samples
Brief Title: Evaluation of the Involvement of the Intestinal Microbiota and Choline Deficiency in the Severity of Chronic Liver Disease Explored by Analyzing Collection of Biological Samples (MICRONACH)
Acronym: MICRONACH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD020-15
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Liver Disease (Alcoholic or Not)
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic liver diseases are common and the two main causes in France are NAFLD (No Alcoholic Fatty Liver Disease Nonalcoholic) and ALD (alcoholic liver disease).

Because of the importance of the current global obesity, NAFLD has become very common and it is estimated that its prevalence in the general population reaches 20-30%.

NAFLD (No Alcoholic Fatty Liver Disease Nonalcoholic) and ALD (alcoholic liver disease) includes a broad spectrum of liver damage, ranging from simple steatosis isolated (infiltration of fat in the liver), in hepatic inflammation, fibrosis (abnormally high accumulation of extracellular components in the functional liver tissue) and finally cirrhosis and its complications.

Choline deficiency (essential nutrient generally classified as Class B vitamins) has been associated with liver damage each characterizing NAFLD and ALD. The amount of choline in the body depends in particular on food intake and degradation of choline by the intestinal microbiota.

NAFLD and ALD are complex pathologies resulting from the interaction of environmental / nutritional factors and a genetic background. It therefore appears now necessary to study the influence of the relationship between genetic predisposition, environmental factors, and gut microbiota metabolism of choline on the severity of liver injury observed in NAFLD and ALD.

If the interaction of these three elements (the host genetics - environmental factors - and intestinal microbiota metabolic choline) has an influence on the severity of the lesions of NAFLD and ALD direct application may be of bring a food supplement choline in patients at risk (mutation of the PEMT gene (phosphatidylethanolamine N-methyltransferase), postmenopausal women, microbiota profile for increased degradation of dietary choline) to restore the amount of choline in the body and thus to avoid a worsening of the ALD or NAFLD and progression to cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD (No alcoholic liver disease) and / or ALD (alcoholic liver disease)
* Liver biopsy scheduled
* NAFLD is defined by the presence of hepatic steatosis (ultrasound or retrospectively confirmed histologically) without concomitant treatment responsible for steatosis (corticosteroids, amiodarone, methotrexate, tamoxifen) without risk drinking of alcoholic beverages (> 210 g / week in men or> 140 g / week in women), and no other cause of chronic liver disease.
* ALD will be defined by the presence of chronic liver disease in a patient with a risk of alcohol consumption (> 210 g / week in men or> 140 g / week in women).
* Obtaining the opposition not to participate in the study
* Obtaining the signature of consent on the collection of biological samples of each participating centers
* Affiliation to the social security system

Exclusion Criteria:

* Cause concomitant chronic liver disease other than NAFLD or ALD
* concomitant treatment responsible for steatosis (steroids, amiodarone, methotrexate, tamoxifen)
* Previous history of bariatric surgery
* Antibiotic treatment in the two months prior to inclusion
* Refusal to participate and / or Non-obtaining consent for collection of biological samples
* Pregnant woman, parturient or nursing mothers. The absence of pregnancy will be provided on condition of effective contraception or after control negativity biological markers of pregnancy (b-HCG)
* Minor Person
* Major Persons subject to enhanced protection, deprived of their liberty by judicial or administrative decision, without consent hospitalized or admitted to a health or social establishment for purposes other than research
* Person who is not affiliated to a social security scheme or of such a regime

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this study will be selected by the investigators of each center among patients for whom a liver biopsy is provided in the clinical management in their center.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with a significant hepatic fibrosis confirmed by a liver biopsy | at baseline (Day of liver biopsy)
  Number of participants with a significant hepatic fibrosis confirmed by a liver biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu SCHNEE, PH, Study Director — CHD Vendée de la Roche sur Yon
Locations (4):
- France (4):
  - CHU Angers, Angers
  - CHU Nantes, Nantes
  - CHU Rennes, Rennes
  - CHU Toulouse, Toulouse